CLINICAL TRIAL: NCT05763576
Title: A Phase I Study to Investigate Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of RO7565020 in Healthy Participants and in Participants With Chronic Hepatitis B Virus Infection
Brief Title: A Study to Investigate Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of RO7565020 in Healthy Participants and in Participants With Chronic Hepatitis B Virus Infection
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: The Sponsor decided to discontinue the development of RO7565020 and as a result the BP44118 study was terminated.
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: BP44118; EU Trial Number (Registry Identifier: 2022-502579-46-00)
Record Dates: First submitted 2023-02-28; First posted 2023-03-10 (Actual); Results first posted 2026-01-22 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Chronic Hepatitis B
MeSH Terms: conditions — Hepatitis B, Chronic | interventions — Nucleobindins; Therapeutics

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- RO7565020 (Experimental)
  Interventions: Drug: RO7565020; Drug: Nucleos(t)ide analogue (NUC) treatment
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: RO7565020 — RO7565020 will be administered by subcutaneous injection or intravenous infusion.
  Arms: RO7565020
Other: Placebo — Matching placebo will be administered by subcutaneous injection or intravenous infusion.
  Arms: Placebo
Drug: Nucleos(t)ide analogue (NUC) treatment — NUC treatment, including tenofovir disoproxil fumarate (TDF), tenofovir alafenamide (TAF), or entecavir (ETV), will be administered orally per local prescribing information.
  Arms: RO7565020

SUMMARY:
This is a first in human (FIH), multi-center, dose-finding, and dose-escalation Phase I clinical study of RO7565020 to investigate the safety and tolerability and to characterize the pharmacokinetics and pharmacodynamics following single and/or multiple doses of RO7565020 in healthy participants and/or virologically suppressed participants with chronic hepatitis B (CHB).

ELIGIBILITY:
Inclusion Criteria:

Healthy volunteers:

* Healthy participants
* Body mass index (BMI) between 18 and 32 kg/m^2

CHB participants:

* CHB infection (HBsAg-positive for >/= 6 months)
* On NUC (ETV, TAF, or TDF) monotherapy for >/= 12 months
* Liver biopsy, FibroScan, or equivalent test within the past 6 months demonstrating liver disease consistent with chronic HBV infection without evidence of bridging fibrosis or cirrhosis
* BMI between 18 and 32 kg/m^2

Exclusion Criteria:

Healthy volunteers:

* History of any clinically significant disease
* Concomitant disease that could interfere with treatment or conduct of study
* Use of any treatment within the 2 weeks or within 5 half-lives prior to first dosing (whichever is longer)

CHB participants:

* Evidence of liver cirrhosis or decompensated liver disease
* History or suspicion of hepatocellular carcinoma (HCC)
* History or evidence of a medical condition associated with chronic liver disease other than HBV infection, or clinically significant and not adequately controlled non-hepatic disease
* History of or currently receiving any systemic anti-neoplastic or immune-modulatory treatment within the 8 weeks prior to the first dosing or the expectation that such treatment will be needed at any time during the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2023-04-28 (Actual); Primary Completion 2024-12-23 (Actual); Study Completion 2024-12-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (9):
- Quest Clinical Research, San Francisco, California, United States
- Hong Kong (2):
  - Queen Mary Hospital, Hong Kong
  - Prince of Wales Hospital, Shatin, New Territories
- New Zealand Clinical Research - Auckland, Auckland, New Zealand
- Hallym University Chuncheon Sacred Heart Hospital, Chuncheon, South Korea
- Hospital Alvaro Cunqueiro, Vigo, Pontevedra, Spain
- Chang Gung Medical Foundation Linkou Branch, Taoyuan, Taiwan
- Thailand (2):
  - Faculty of Medicine Siriraj Hospital, Bangkok
  - Maharaj Nakorn Chiang Mai Hospital, Chiang Mai

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 48 healthy participants (Part 1a) and 12 participants with chronic hepatitis B (CHB) virus infection (Part 2a) took part in the study across 10 investigative sites in Hong Kong, Thailand, New Zealand, Republic of Korea, United States, Spain, and Taiwan from 28 April 2023 to 23 December 2024.
Pre-assignment Details: The study consists of 3 parts- Part 1a: single-ascending dose (SAD) and Part 1b: multiple doses in healthy participants, Part 2 (a and b): SAD in participants with CHB, and Part 3: multiple doses in participants with CHB. No participants were enrolled in the Part 1b, Part 2b, and Part 3 as the study was terminated by the sponsor.
Groups:
- Part 1a Placebo: Healthy participants received a single dose of placebo, matched to each dose level of RO7565020, via subcutaneous (SC) injection or intravenous (IV) infusion on Day 1 of treatment period.
- Part 1a Cohort 1: Healthy participants received a single dose of RO7565020, 70 milligrams (mg) as a SC injection on Day 1 of treatment period.
- Part 1a Cohort 2: Healthy participants received a single dose of RO7565020, 230 mg as a SC injection on Day 1 of treatment period.
- Part 1a Cohort 3: Healthy participants received a single dose of RO7565020, 360 mg as a SC injection on Day 1 of treatment period.
- Part 1a Cohort 4: Healthy participants received a single dose of RO7565020, 360 mg as an IV infusion on Day 1 of treatment period.
- Part 1a Cohort 5: Healthy participants received a single dose of RO7565020, 1500 mg as an IV infusion on Day 1 of treatment period.
- Part 1a Cohort 6: Healthy participants received a single dose of RO7565020, 360 mg as an SC injection on Day 1 of treatment period. Cohort 6 was a pharmacokinetic (PK) ethnicity bridging cohort between a global population and Chinese population.
- Part 2a Cohort 1: Participants with CHB who were virologically suppressed with stable nucleos(t)ide analogue (NUC) treatment received a single dose of RO7565020, 70 mg, as an SC injection on Day 1 of treatment period.
- Part 2a Cohort 2: Participants with CHB who were virologically suppressed with stable NUC treatment received a single dose of RO7565020, 230 mg, as an SC injection on Day 1 of treatment period.
Period: Overall Study
Arm/Group | Part 1a Placebo | Part 1a Cohort 1 | Part 1a Cohort 2 | Part 1a Cohort 3 | Part 1a Cohort 4 | Part 1a Cohort 5 | Part 1a Cohort 6 | Part 2a Cohort 1 | Part 2a Cohort 2
Started | 12 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6
Completed | 12 | 6 | 6 | 6 | 6 | 5 | 6 | 4 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 6
Not completed — Study Terminated by Sponsor | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 6
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety population included all participants randomized/assigned to study treatment and who received at least one dose of the study treatment, whether prematurely withdrawn from the study or not.
Groups:
- Part 1a Placebo: Healthy participants received a single dose of placebo, matched to each dose level of RO7565020, via SC injection or IV infusion on Day 1 of treatment period.
- Part 1a Cohort 1: Healthy participants received a single dose of RO7565020, 70 mg as a SC injection on Day 1 of treatment period.
- Part 1a Cohort 6: Healthy participants received a single dose of RO7565020, 360 mg as an SC injection on Day 1 of treatment period. Cohort 6 was a PK ethnicity bridging cohort between a global population and Chinese population.
- Part 2a Cohort 1: Participants with CHB who were virologically suppressed with stable NUC treatment received a single dose of RO7565020, 70 mg, as an SC injection on Day 1 of treatment period.
- Total: Total of all reporting groups
Arm/Group | Part 1a Placebo | Part 1a Cohort 1 | Part 1a Cohort 2 | Part 1a Cohort 3 | Part 1a Cohort 4 | Part 1a Cohort 5 | Part 1a Cohort 6 | Part 2a Cohort 1 | Part 2a Cohort 2 | Total
Number analyzed (Participants) | 12 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 60
Age, Continuous [Mean (Standard Deviation); unit: years] | 34.2 (9.3) | 39.8 (7.9) | 34.8 (12.4) | 47.3 (8.6) | 39.0 (13.1) | 38.5 (11.2) | 35.7 (10.6) | 52.8 (4.4) | 48.7 (8.2) | 40.5 (11.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 3 | 5 | 1 | 2 | 4 | 0 | 1 | 1 | 23
  Male | 6 | 3 | 1 | 5 | 4 | 2 | 6 | 5 | 5 | 37
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 3
  Not Hispanic or Latino | 11 | 5 | 6 | 6 | 6 | 5 | 6 | 6 | 5 | 56
  Unknown or Not Reported | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 4 | 0 | 1 | 1 | 2 | 1 | 6 | 6 | 5 | 26
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 2
  Black or African American | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  White | 4 | 5 | 4 | 5 | 3 | 4 | 0 | 0 | 1 | 26
  More than one race | 2 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 4
  Unknown or Not Reported | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Part 1a: Number of Healthy Volunteers With Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: An AE was any untoward medical occurrence in a participant administered a pharmaceutical product and which does not necessarily have to have a causal relationship with the treatment. An AE can therefore be any unfavorable and unintended sign (including abnormal laboratory finding), symptoms, or disease temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. SAE is any significant hazard, contraindication, or side effect that is fatal or life-threatening, requires hospitalization or prolongation of an existing hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect, is medically significant or requires intervention.
Time Frame: Up to approximately 40 weeks
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Groups:
- Part 1a Cohort 6: Healthy participants received a single dose of RO7565020, 360 mg as a SC injection on Day 1 of treatment period. Cohort 6 was a PK ethnicity bridging cohort between a global population and Chinese population.
Arm/Group | Part 1a Placebo | Part 1a Cohort 1 | Part 1a Cohort 2 | Part 1a Cohort 3 | Part 1a Cohort 4 | Part 1a Cohort 5 | Part 1a Cohort 6
Number analyzed (Participants) | 12 | 6 | 6 | 6 | 6 | 6 | 6
Participants
  AEs | 6 | 4 | 5 | 4 | 6 | 6 | 1
  SAEs | 0 | 0 | 0 | 0 | 1 | 0 | 0

2. Primary Outcome: Part 2a: Number of CHB Participants With AEs and SAEs
Description: as for outcome 1
Time Frame: Up to approximately 32 weeks
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Groups:
- Part 2a Cohort 1: Participants with CHB who were virologically suppressed with stable NUC treatment received a single dose of RO7565020, 70 mg, as a SC injection on Day 1 of treatment period.
- Part 2a Cohort 2: Participants with CHB who were virologically suppressed with stable NUC treatment received a single dose of RO7565020, 230 mg, as a SC injection on Day 1 of treatment period.
Arm/Group | Part 2a Cohort 1 | Part 2a Cohort 2
Number analyzed (Participants) | 6 | 6
Participants
  AEs | 2 | 3
  SAEs | 0 | 0

3. Primary Outcome: Part 1a: Number of Healthy Volunteers With Adverse Events of Special Interest (AESI)
Description: An AE was any untoward medical occurrence in a participant administered a pharmaceutical product and which does not necessarily have to have a causal relationship with the treatment. An AE can therefore be any unfavorable and unintended sign (including abnormal laboratory finding), symptoms, or disease temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. AESI includes elevated alanine aminotransferase (ALT) or aspartate aminotransferase (AST) value in combination with either an elevated bilirubin value or clinical jaundice and suspected transmission of an infectious agent by the study treatment.
Time Frame: Up to approximately 40 weeks
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1a Placebo | Part 1a Cohort 1 | Part 1a Cohort 2 | Part 1a Cohort 3 | Part 1a Cohort 4 | Part 1a Cohort 5 | Part 1a Cohort 6
Number analyzed (Participants) | 12 | 6 | 6 | 6 | 6 | 6 | 6
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0

4. Primary Outcome: Part 2a: Number of CHB Participants With AESI
Description: An AE was any untoward medical occurrence in a participant administered a pharmaceutical product and which does not necessarily have to have a causal relationship with the treatment. An AE can therefore be any unfavorable and unintended sign (including abnormal laboratory finding), symptoms, or disease temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. AESI includes elevated ALT or AST value in combination with either an elevated bilirubin value or clinical jaundice and suspected transmission of an infectious agent by the study treatment.
Time Frame: Up to approximately 32 weeks
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2a Cohort 1 | Part 2a Cohort 2
Number analyzed (Participants) | 6 | 6
Participants | 0 | 0

5. Secondary Outcome: Part 1a (SC Cohorts) and Part 2a: Time to Maximum Concentration (Tmax) of RO7565020
Time Frame: Part 1a: Predose, 1, 4, and 8 hours post-dose on Day 1; Days 2, 3, 4, 8, 15, 21, 29, 57, 85, 141, 197, and 253. Part 2a: Predose, 1, 4, and 8 hours post-dose on Day 1; Days 2, 3, 4, 8, 15, 22, 29, 57, 85, 113, 141, and 169
Population: PK-evaluable population included all participants who received at least one dose of study treatment and who had data from at least one postdose sample. Overall number analyzed is the number of participants with data available for analysis.
Measure: Median (Full Range); unit: day
Arm/Group | Part 1a Cohort 1 | Part 1a Cohort 2 | Part 1a Cohort 3 | Part 1a Cohort 6 | Part 2a Cohort 1 | Part 2a Cohort 2
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 5 | 6
day | 14 [2 to 56] | 17 [6.99 to 21] | 10.5 [3 to 28] | 10.7 [6.06 to 29.1] | 7.01 [3.03 to 21] | 10.5 [6.96 to 15]

6. Secondary Outcome: Part 1a (IV Cohorts): Tmax of RO7565020
Time Frame: Predose, 0.08, 1, 4, and 8 hours post-dose on Day 1; Days 2, 3, 4, 8, 15, 21, 29, 57, 85, 141, 197, and 253
Population: PK-evaluable population included all participants who received at least one dose of study treatment and who had data from at least one postdose sample.
Measure: Median (Full Range); unit: hours
Arm/Group | Part 1a Cohort 4 | Part 1a Cohort 5
Number analyzed (Participants) | 6 | 6
hours | 2.12 [2.12 to 6.3] | 2.12 [2.12 to 2.17]

7. Secondary Outcome: Parts 1a and 2a: Maximum Serum Concentration (Cmax) of RO7565020
Time Frame: Both Part 1a & 2a Cohorts: Predose, 1, 4, 8 hours post-dose on Day 1; Days 2, 3, 4, 8, 15, 29, 57, 85, & 141. Additionally, Part 1a: Days 21, 197, & 253; Part 2a: Days 22, 113, & 169; IV Cohorts: 0.08 hours after start of infusion, Days 21, 197, & 253
Population: as for outcome 5
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: micrograms per milliliter (μg/mL)
Arm/Group | Part 1a Cohort 1 | Part 1a Cohort 2 | Part 1a Cohort 3 | Part 1a Cohort 4 | Part 1a Cohort 5 | Part 1a Cohort 6 | Part 2a Cohort 1 | Part 2a Cohort 2
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 5 | 6
micrograms per milliliter (μg/mL) | 4.99 (52.1) | 14.4 (66.0) | 29.4 (37.1) | 165 (18.6) | 587 (27.6) | 27.7 (43.3) | 2.96 (46.5) | 18.2 (45.7)

8. Secondary Outcome: Parts 1a and 2a: Area Under the Time-concentration Curve From Time 0 to Time of Last Sampling Point or Last Quantifiable Sample, Whichever Comes First (AUC0-last) of RO7565020
Time Frame: as for outcome 7
Population: as for outcome 6
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: day*μg/mL
Arm/Group | Part 1a Cohort 1 | Part 1a Cohort 2 | Part 1a Cohort 3 | Part 1a Cohort 4 | Part 1a Cohort 5 | Part 1a Cohort 6 | Part 2a Cohort 1 | Part 2a Cohort 2
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6
day*μg/mL | 559 (42.0) | 1630 (50.0) | 3390 (33.8) | 6630 (19.6) | 24800 (17.0) | 2960 (33.4) | 59.9 (575.4) | 898 (121.2)

9. Secondary Outcome: Parts 1a and 2a: Area Under the Time-concentration Curve From Time 0 to Infinity (AUC0-inf) of RO7565020
Time Frame: as for outcome 7
Population: as for outcome 5
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: day*μg/mL
Arm/Group | Part 1a Cohort 1 | Part 1a Cohort 2 | Part 1a Cohort 3 | Part 1a Cohort 4 | Part 1a Cohort 5 | Part 1a Cohort 6 | Part 2a Cohort 1 | Part 2a Cohort 2
Number analyzed (Participants) | 6 | 1 | 4 | 2 | 2 | 3 | 3 | 4
day*μg/mL | NA (NA) — Geometric mean (GM) and Geometric coefficient of variation were not available because, based on Roche internal non-compartmental analysis (NCA) guiding principles (version 4.0), these could only be provided when the terminal phase constant (lambda_z) was appropriately determined and/or the extrapolated percentage of AUC0-inf was less than 20%. Data is not available as neither of these conditions were met for this cohort. | 2180 (NA) — Geometric coefficient of variation was not estimable for one participant. | 3660 (24.4) | 8450 (10.2) | 30700 (26.7) | 2900 (25.7) | 172 (45.3) | 792 (183.9)

10. Secondary Outcome: Parts 1a and 2a: Terminal Half-life (t1/2) of RO7565020
Time Frame: as for outcome 7
Population: as for outcome 5
Measure: Median (Full Range); unit: day
Arm/Group | Part 1a Cohort 1 | Part 1a Cohort 2 | Part 1a Cohort 3 | Part 1a Cohort 4 | Part 1a Cohort 5 | Part 1a Cohort 6 | Part 2a Cohort 1 | Part 2a Cohort 2
Number analyzed (Participants) | 6 | 1 | 4 | 2 | 2 | 3 | 3 | 4
day | NA [NA to NA] — Median and full range were not available because, based on Roche internal NCA guiding principles (version 4.0), these could only be provided when the terminal phase constant (lambda_z) was appropriately determined and/or the extrapolated percentage of AUC0-inf was less than 20%. Data is not available as neither of these conditions were met for this cohort. | 88 [88 to 88] | 88.3 [80.1 to 92.3] | 83.3 [80.4 to 86.2] | 94.8 [88.9 to 101] | 78.2 [71.6 to 86.2] | 13.6 [4.69 to 29.6] | 19.8 [4.8 to 51.7]

11. Secondary Outcome: Part 1a (IV Cohorts): Volume of Distribution (Vss) of RO7565020
Time Frame: Predose, 0.08, 1, 4, and 8 hours post-dose on Day 1; Days 2, 3, 4, 8, 15, 21, 29, 57, 85, 141, 197 and 253
Population: as for outcome 5
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: liters
Arm/Group | Part 1a Cohort 4 | Part 1a Cohort 5
Number analyzed (Participants) | 2 | 2
liters | 5.14 (2.5) | 6.19 (37.3)

12. Secondary Outcome: Part 1a (IV Cohorts): Clearance (CL) of RO7565020
Time Frame: Predose, 0.08, 1, 4, and 8 hours post-dose on Day 1; Days 2, 3, 4, 8, 15, 21, 29, 57, 85, 141, 197 and 253
Population: as for outcome 5
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: milliliter/hour (mL/h)
Arm/Group | Part 1a Cohort 4 | Part 1a Cohort 5
Number analyzed (Participants) | 2 | 2
milliliter/hour (mL/h) | 1.78 (10.2) | 2.03 (26.7)

13. Secondary Outcome: Part 1a (SC Cohorts) and Part 2a: Apparent Clearance (CL/F) of RO7565020
Time Frame: as for outcome 5
Population: as for outcome 5
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mL/h
Arm/Group | Part 1a Cohort 1 | Part 1a Cohort 2 | Part 1a Cohort 3 | Part 1a Cohort 6 | Part 2a Cohort 1 | Part 2a Cohort 2
Number analyzed (Participants) | 6 | 1 | 4 | 3 | 3 | 4
mL/h | NA (NA) — GM and Geometric coefficient of variation were not available because, based on Roche internal NCA guiding principles (version 4.0), these could only be provided when the terminal phase constant (lambda_z) was appropriately determined and/or the extrapolated percentage of AUC0-inf was less than 20%. Data is not available as neither of these conditions were met for this cohort. | 4.39 (NA) — Geometric coefficient of variation was not estimable for one participant. | 4.1 (24.4) | 5.18 (25.7) | 16.9 (45.3) | 12.1 (183.9)

14. Secondary Outcome: Part 1a (SC Cohorts) and Part 2a: Apparent Volume of Distribution (Vz/F) at Terminal Phase of RO7565020
Time Frame: as for outcome 5
Population: as for outcome 5
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: liters
Arm/Group | Part 1a Cohort 1 | Part 1a Cohort 2 | Part 1a Cohort 3 | Part 1a Cohort 6 | Part 2a Cohort 1 | Part 2a Cohort 2
Number analyzed (Participants) | 6 | 1 | 4 | 3 | 3 | 4
liters | NA (NA) — GM and Geometric coefficient of variation were not available because, based on Roche internal NCA guiding principles (version 4.0), these could only be provided when the terminal phase constant (lambda_z) was appropriately determined and/or the extrapolated percentage of AUC0-inf was less than 20%. Data is not available as neither of these conditions were met for this cohort. | 13.4 (NA) — Geometric coefficient of variation was not estimable for one participant. | 12.4 (26.8) | 14.1 (18.3) | 7.23 (60.8) | 7.33 (35.0)

15. Secondary Outcome: Part 2a: Change From Baseline in Serum Quantitative Hepatitis B Surface Antigen (HBsAg)
Description: IU/mL= international units per milliliter
Time Frame: Baseline, 4- and 8-hours post-dose on Day 1; subsequently on Days 2, 3, 4, 8, 15, 22, 29, 57, 85, 113, 141, and 169
Population: Pharmacodynamic (PD) population included all participants with CHB who received at least one dose of study treatment. Number analyzed is the number of participants with data available for analysis at the specified timepoint.
Measure: Mean (Standard Deviation); unit: log10 IU/mL
Arm/Group | Part 2a Cohort 1 | Part 2a Cohort 2
Number analyzed (Participants) | 6 | 6
log10 IU/mL
  Baseline | 2.36 (0.73) | 2.63 (0.38)
  Change at 4 h Post-dose, Day 1 | -0.20 (0.09) | -0.63 (0.45)
  Change at 8 h Post-dose, Day 1 | -0.44 (0.24) | -0.96 (0.39)
  Change at Day 2 | -0.88 (0.29) | -1.03 (0.33)
  Change at Day 3 | -0.99 (0.29) | -1.12 (0.28)
  Change at Day 4 | -1.03 (0.29) | -1.10 (0.27)
  Change at Day 8: number analyzed (Participants) | 5 | 6
  Change at Day 8 | -1.38 (0.54) | -1.43 (0.29)
  Change at Day 15: number analyzed (Participants) | 5 | 6
  Change at Day 15 | -1.17 (0.56) | -1.29 (0.26)
  Change at Day 22: number analyzed (Participants) | 5 | 6
  Change at Day 22 | -1.04 (0.58) | -1.19 (0.25)
  Change at Day 29: number analyzed (Participants) | 5 | 6
  Change at Day 29 | -1.01 (0.57) | -1.16 (0.27)
  Change at Day 57: number analyzed (Participants) | 5 | 6
  Change at Day 57 | -0.68 (0.60) | -1.06 (0.39)
  Change at Day 85 | -0.51 (0.57) | -0.87 (0.55)
  Change at Day 113: number analyzed (Participants) | 5 | 0
  Change at Day 113 | -0.58 (0.56) |
  Change at Day 141: number analyzed (Participants) | 5 | 0
  Change at Day 141 | -0.54 (0.53) |
  Change at Day 169 | -0.29 (0.56) | -0.48 (0.67)

16. Secondary Outcome: Part 2a: Maximum Reduction From Baseline in Serum HBsAg
Time Frame: Up to Day 169
Population: PD population included all participants with CHB who received at least one dose of study treatment.
Measure: Mean (Standard Deviation); unit: log10 IU/mL
Arm/Group | Part 2a Cohort 1 | Part 2a Cohort 2
Number analyzed (Participants) | 6 | 6
log10 IU/mL | -1.39 (0.471) | -1.44 (0.288)

17. Secondary Outcome: Part 2a: Percentage of Participants With HBsAg Loss
Time Frame: Up to Day 169
Population: PD population included all participants with CHB who received at least one dose of study treatment.
Measure: Number; unit: percentage of participants
Arm/Group | Part 2a Cohort 1 | Part 2a Cohort 2
Number analyzed (Participants) | 6 | 6
percentage of participants | 0 | 0

18. Secondary Outcome: Part 2a: Percentage of Participants With HBsAg Seroconversion
Description: HBsAg seroconversion was defined as sustained loss of HBsAg and detection of anti-HBs antibody.
Time Frame: Up to Day 169
Population: PD population included all participants with CHB who received at least one dose of study treatment.
Measure: Number; unit: percentage of participants
Arm/Group | Part 2a Cohort 1 | Part 2a Cohort 2
Number analyzed (Participants) | 6 | 6
percentage of participants | 0 | 0

19. Secondary Outcome: Part 2a: Percentage of Participants With Hepatitis B e Antigen (HBeAg) Loss Among HBeAg-positive Participants at Baseline
Time Frame: At Days 2, 3, 4, 8, 15, 22, 29, 57, 85, 113, 141, and 169
Population: PD population included all participants with CHB who received at least one dose of study treatment. Overall Number analyzed included participants who were HBeAg-positive at baseline.
Measure: Number; unit: percentage of participants
Arm/Group | Part 2a Cohort 1 | Part 2a Cohort 2
Number analyzed (Participants) | 1 | 2
percentage of participants
  Day 2 | 0 | 0
  Day 3 | 0 | 0
  Day 4 | 0 | 0
  Day 8 | 0 | 50.0
  Day 15 | 0 | 50.0
  Day 22 | 0 | 50.0
  Day 29 | 0 | 50.0
  Day 57 | 0 | 50.0
  Day 85 | 0 | 0
  Day 113 | 0 | 0
  Day 141 | 0 | 0
  Day 169 | 0 | 50.0

20. Secondary Outcome: Part 2a: Percentage of Participants With HBeAg Seroconversion Among HBeAg-positive Participants at Baseline
Description: HBeAg seroconversion was defined as sustained loss of HBeAg and detection of anti-HBe antibody.
Time Frame: Up to Day 169
Population: as for outcome 19
Measure: Number; unit: percentage of participants
Arm/Group | Part 2a Cohort 1 | Part 2a Cohort 2
Number analyzed (Participants) | 1 | 2
percentage of participants | 0 | 0

21. Secondary Outcome: Number of Participants With Anti-Drug Antibodies (ADAs) to RO7565020
Description: The number of ADA-positive participants at baseline (baseline prevalence) and after drug administration was determined in participants exposed to RO7565020 (post-baseline). Participants were considered ADA positive if they had ADA negative or have missing data at baseline but develop an ADA response following study treatment administration (treatment-induced ADA response), or if they are ADA positive at baseline and the titer of one or more post-baseline samples is at least 4-fold (e.g., ≥ 0.60-titer units) greater than the titer of the baseline sample (treatment enhanced ADA response).
Time Frame: Part 1a: Baseline and post-baseline (up to approximately 40 weeks); Part 2a: Baseline and post-baseline (up to approximately 32 weeks)
Population: Immunogenicity population included participants who had at least one ADA assessment and analyzed according to the treatment they actually received. Number analyzed is the number of participants with data available for analysis at the specified timepoint.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1a Placebo | Part 1a Cohort 1 | Part 1a Cohort 2 | Part 1a Cohort 3 | Part 1a Cohort 4 | Part 1a Cohort 5 | Part 1a Cohort 6 | Part 2a Cohort 1 | Part 2a Cohort 2
Number analyzed (Participants) | 12 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6
Participants
  Baseline | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Post-baseline: number analyzed (Participants) | 0 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6
  Post-baseline | 0 | 0 | 2 | 0 | 3 | 1 | 4 | 1 | 0

ADVERSE EVENTS:
Time Frame: Part 1a: Up to approximately 40 weeks Part 2a: Up to approximately 32 weeks
Description: Safety population included all participants randomized/assigned to study treatment and who received at least one dose of the study treatment, whether prematurely withdrawn from the study or not.
Arm/Group | Part 1a Placebo | Part 1a Cohort 1 | Part 1a Cohort 2 | Part 1a Cohort 3 | Part 1a Cohort 4 | Part 1a Cohort 5 | Part 1a Cohort 6 | Part 2a Cohort 1 | Part 2a Cohort 2
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/6 | 0/6 | 0/6 | 1/6 | 0/6 | 0/6 | 0/6 | 0/6
Other Adverse Events (participants affected / at risk) | 6/12 | 4/6 | 5/6 | 4/6 | 6/6 | 6/6 | 1/6 | 2/6 | 3/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part 1a Placebo (N=12) | Part 1a Cohort 1 (N=6) | Part 1a Cohort 2 (N=6) | Part 1a Cohort 3 (N=6) | Part 1a Cohort 4 (N=6) | Part 1a Cohort 5 (N=6) | Part 1a Cohort 6 (N=6) | Part 2a Cohort 1 (N=6) | Part 2a Cohort 2 (N=6)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part 1a Placebo (N=12) | Part 1a Cohort 1 (N=6) | Part 1a Cohort 2 (N=6) | Part 1a Cohort 3 (N=6) | Part 1a Cohort 4 (N=6) | Part 1a Cohort 5 (N=6) | Part 1a Cohort 6 (N=6) | Part 2a Cohort 1 (N=6) | Part 2a Cohort 2 (N=6)
Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eustachian tube dysfunction (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoacusis (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cataract (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain lower (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infrequent bowel movements (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Catheter site bruise (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Influenza like illness (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
COVID-19 (Infections and infestations) | 2 (2) | 1 (1) | 2 (2) | 1 (1) | 3 (4) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Conjunctivitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oral herpes (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 2 (3) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Viral upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Arthropod bite (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ligament sprain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin laceration (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 2 (3) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Migraine (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Somnolence (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Endometriosis (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Intermenstrual bleeding (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vaginal discharge (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vaginal haemorrhage (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin striae (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-05-15): https://cdn.clinicaltrials.gov/large-docs/76/NCT05763576/Prot_SAP_000.pdf